CLINICAL TRIAL: NCT01271751
Title: A Pilot Study to Evaluate the Efficacy and Safety of GFT505 (80mg) Orally Administered Once Daily for 28 Days in Atherogenic Dyslipidaemic Patients With Abdominal Obesity. A Double Blind, Placebo-controlled and Randomized Study.
Brief Title: Pilot Study With GFT505 (80mg) in Atherogenic Dyslipidaemic Patients With Abdominal Obesity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genfit (Industry)
Responsible Party: Product Development Department, Genfit
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GFT505-208-3; 2008-005779-86 (EudraCT Number)
Record Dates: First submitted 2011-01-06; First posted 2011-01-07 (Estimated); Last update posted 2011-01-07 (Estimated); Status verified 2011-01

CONDITIONS: Atherogenic Dyslipidaemia; Abdominal Obesity
Keywords: Atherogenic-dyslipidaemia; PPARs
MeSH Terms: conditions — Obesity, Abdominal | interventions — 2-(2,6-dimethyl-4-(3-(4-(methylthio)phenyl)-3-oxo-1-propenyl)phenoxyl)-2-methylpropanoic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GFT505 80mg (Experimental)
  Interventions: Drug: GFT505 80mg
- Matching placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GFT505 80mg — hard gelatin capsules dosed at 20mg, oral administration, 4 capsules per day before breakfast
  Arms: GFT505 80mg
Drug: Placebo — hard gelatin capsules, oral administration, 4 capsules per day before breakfast
  Arms: Matching placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of GFT505 80mg in reducing serum Triglycerides (TG) and increasing High Density Lipoprotein Cholesterol (HDL-C) levels compared with placebo in atherogenic dyslipidaemic patients with abdominal obesity, and to assess the tolerability and safety of once-a-day administrations of oral doses of GFT505 during 28 days.

DETAILED DESCRIPTION:
The study period per patient is 7 to 14 weeks: a screening period (1 to 8 weeks) will precede a 4-week double-blind treatment period and a 2-week follow-up period.

During the screening period, patients will be asked to start or continue adequate diet and exercise and to stop their lipid-lowering medication (for not treatment-naïve patients). For patient taking any lipid-regulating medication, a minimum of 8-week wash-out from lipid-regulating therapies (fibrates, statins, …) is required.

ELIGIBILITY:
Inclusion Criteria:

* Male or post-menopausal female.
* Waist circumference ≥102cm for male, ≥ 88cm for female.
* Atherogenic dislipidaemia inadequately controlled despite Therapeutic Lifestyle Change (TLC) recommendations (diet and exercise).
* 150≤ fasting TG ≤ 600 mg/dL (1.69 ≤ fasting TG ≤ 6.78 mmol/L) at V2.
* Fasting HDL-C ≤ 40 mg/dL (≤ 1.03 mmol/L) for male, HDL-C ≤ 45 mg/dL (≤ 1.16 mmol/L) for female at V2.

Exclusion Criteria:

* Body Mass Index (BMI) ≥ 40 kg/m².
* Blood Pressure > 160 / 95 mmHg.
* Type I or type II Diabetes Mellitus.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2009-01; Primary Completion 2009-09 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Decrease in serum Triglycerides (TG) level | 28 days
  To evaluate the efficacy of GFT505 80mg in reducing serum TG compared with placebo. Evaluation will be made during the selection period, then the first day prior any drug intake, 2 and 4 weeks after the first treatment intake and 2 weeks after the last treatment intake (follow-up visit)
Increase in serum High Density Lipoprotein Cholesterol (HDL-C) level | 28 days
  To evaluate the efficacy of GFT505 80mg in increasing HDL-C levels compared with placebo. Evaluation will be made during the selection period, then the first day prior any drug intake, 2 and 4 weeks after the first treatment intake and 2 weeks after the last treatment intake (follow-up visit)

SECONDARY OUTCOMES:
Decrease in Low Density Lipoprotein Cholesterol (LDL-C) levels | 28 days
  To evaluate the efficacy of GFT505 80mg in reducing LDL-C levels compared with placebo. Evaluation will be made during the selection period, then the first day prior any drug intake, 2 and 4 weeks after the first treatment intake and 2 weeks after the last treatment intake (follow-up visit)
Decrease in non-HDL-C (High Density Lipoprotein Cholesterol) levels | 28 days
  To evaluate the efficacy of GFT505 80mg in reducing non-HDL-C levels compared with placebo. Evaluation will be made during the selection period, then the first day prior any drug intake, 2 and 4 weeks after the first treatment intake and 2 weeks after the last treatment intake (follow-up visit)

CONTACTS AND LOCATIONS:
Overall Officials: Rémy Hanf, Development Director, Study Director — GENFIT, France; Eric BRUCKERT, Pr., Study Chair — University Hospital of Paris 6, France
Locations (47):
- France (36):
  - Site n°36, Aigrefeuille-sur-Maine
  - Site n°78, Angers
  - Site n°79, Angers
  - Site n°80, Angers
  - Site n°82, Angers
  - Site n°21, Bauné
  - Site n°16, Beaucouzé
  - Site n°18, Briollay
  - Site n°14, Cholet
  - Site n°26, Cholet
  - Site n°42, Haute-Goulaine
  - Site n°45, Héric
  - Site n°32, La Chapelle-sur-Erdre
  - Site n°11, La Jubaudière
  - Site n°30, La Montagne
  - Site n°91, Laval
  - Site n°23, Le Mesnil-en-Vallée
  - Site n°35, Le Temple-de-Bretagne
  - Site n°12, Les Ponts-de-Cé
  - Site n°17, Montreuil-Juigné
  - Site n°74, Montrevault
  - Site n°10, Murs-Erigné
  - Site n°19, Murs-Erigné
  - Site n°40, Nantes
  - Site n°37, Nantes
  - Site n°31, Nantes
  - Site n°34, Nantes
  - Site n°41, Nort-sur-Erdre
  - Site n°33, Orvault
  - Site n°1, Paris
  - Site n°38, Saint-Étienne-de-Montluc
  - Site n°39, Sautron
  - Site n°13, Segré
  - Site n°75, Tiercé
  - Site n°77, Tiercé
  - Site n°20, Vihiers
- Romania (6):
  - Site n°64, Brasov
  - Site n°61, Bucharest
  - Site n°60, Bucharest
  - Site n°63, Bucharest
  - Site n°62, Bucharest
  - Site n°65, Craiova
- Tunisia (5):
  - Site n°52, Bab Sâadoun Tunis
  - Site n°53, Bab Sâadoun Tunis
  - Site n°50, Tunis
  - Site n°51, Tunis
  - Site n°55, Tunis

REFERENCES:
- [Derived] Staels B, Rubenstrunk A, Noel B, Rigou G, Delataille P, Millatt LJ, Baron M, Lucas A, Tailleux A, Hum DW, Ratziu V, Cariou B, Hanf R. Hepatoprotective effects of the dual peroxisome proliferator-activated receptor alpha/delta agonist, GFT505, in rodent models of nonalcoholic fatty liver disease/nonalcoholic steatohepatitis. Hepatology. 2013 Dec;58(6):1941-52. doi: 10.1002/hep.26461. Epub 2013 Oct 29. PMID 23703580
- [Derived] Cariou B, Zair Y, Staels B, Bruckert E. Effects of the new dual PPAR alpha/delta agonist GFT505 on lipid and glucose homeostasis in abdominally obese patients with combined dyslipidemia or impaired glucose metabolism. Diabetes Care. 2011 Sep;34(9):2008-14. doi: 10.2337/dc11-0093. Epub 2011 Aug 4. PMID 21816979